CLINICAL TRIAL: NCT04171817
Title: Clinical Trial of a Disinfectant Intervention in Therapy Dogs to Combat Hospital-associated Pathogens and Promote Sustainability of Animal-Assisted Visitation Programs
Brief Title: Animal-Assisted Visitation Program Chlorhexidine Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Children's Hospital of Philadelphia (Other); University of Pennsylvania (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01HD097692 (NIH); IRB00205311 (Other: JHM IRB)
Record Dates: First submitted 2019-11-14; First posted 2019-11-21 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Methicillin-resistant Staphylococcus Aureus; Clostridium Difficile; Pseudomonas Aeruginosa
Keywords: therapy dog; canine; animal assisted intervention; chlorhexidine; child
MeSH Terms: conditions — Pseudomonas Infections | interventions — Chlorhexidine

STUDY DESIGN:
Intervention Model Description: This is a multicenter, parallel-arm randomized controlled trial, with 1:1 allocation for intervention versus control. Among those randomized to intervention, dog-handler teams will be additionally randomized to Intervention A first, with crossover to Intervention B, or to Intervention B first, with crossover to Intervention A.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): Dog-handler teams will follow established hospital and therapy dog program guidelines for infection control with no changes for eight sessions. Participants enrolled in the session will derive their Arm assignment from the dog-handler team with which they interact.
- CHX Intervention A (Experimental): Dog-handler teams will follow a modified protocol for infection control, with Treatment A first for four sessions, and cross-over to Treatment B for four sessions. Participants enrolled in the session will derive their Arm assignment from the dog-handler team with which they interact.
  Treatment A consists of a pre-session shampoo with a commercial veterinary chlorhexidine-based product (2-4% chlorhexidine) within 24 hours prior to the session, and wiping with a chlorhexidine-impregnated cloth (2-4% chlorhexidine) at arrival at the session and every 20 minutes during the session, or between participants if the flow of participants is structured in a way that allows this (such as visits from one room to the next to visit individual patients).
  Interventions: Drug: Chlorhexidine
- CHX Intervention B (Experimental): Dog-handler teams will follow a modified protocol for infection control, with Treatment B first for four sessions, and cross-over to Treatment A for four sessions. Participants enrolled in the session will derive their Arm assignment from the dog-handler team with which they interact.
  Treatment B will consist of the same pre-session shampoo with a commercial veterinary chlorhexidine-based product (2-4% chlorhexidine), with a single wipe with a chlorhexidine-impregnated cloth (2-4% chlorhexidine) at arrival. This treatment will depend on the residual activity of chlorhexidine throughout the visit.
  Interventions: Drug: Chlorhexidine

INTERVENTIONS:
Drug: Chlorhexidine — The goal of this work is to assess the effect of chlorhexidine (CHX)-based interventions--specifically use of pre-session chlorhexidine shampoo for the dog and use of chlorhexidine wipes on the dog's fur--on patient exposure to hospital-associated pathogens during the sessions with the dogs
  Other Names: CHX
  Arms: CHX Intervention A; CHX Intervention B

SUMMARY:
Hospital-based Animal-Assisted visitation programs are important complementary therapies, but concerns with infection control may challenge the sustainability of these programs. Pilot data suggest that a low-cost chlorhexidine-based intervention targeted to the dogs involved in the visitation programs holds high potential to prevent pathogen transmission during sessions. In this study, the following aims will be tested: 1) To identify program-related risk factors for acquisition of hospital-associated pathogens by pediatric patients during animal-assisted intervention (AAI) sessions during an initial run-in phase of no intervention; 2) To determine the effect of chlorhexidine (CHX)-based interventions on acquisition of hospital-associated pathogens and microbial communities by patients during AAI sessions via a multicenter randomized controlled trial; and 3) To determine whether the specific benefits achieved by the visitation program, i.e. reduction in blood pressure, heart rate and self-reported pain and anxiety, are impacted by the interventions.

DETAILED DESCRIPTION:
Hospital-based Animal-Assisted visitation programs provide an important complementary treatment in holistic patient care and reduce patient stress, pain and anxiety. However, the risk of transmission of pathogens, such as methicillin-resistant Staphylococcus aureus, is a challenge to the sustainability of hospital-based Animal-Assisted visitation programs. Pilot data suggest that a low-cost chlorhexidine-based intervention targeted to the dogs involved in the visitation programs holds high potential to prevent pathogen transmission during sessions. Therefore, child participants will be enrolled who interact with 40 dogs over twelve sessions (four observational, eight where the dog is randomized to intervention or control) at two enrollment centers. The following aims will be tested: 1) To identify program-related risk factors for acquisition of hospital-associated pathogens by pediatric patients during animal-assisted intervention (AAI) sessions during an initial run-in phase of no intervention; 2) To determine the effect of chlorhexidine (CHX)-based interventions on acquisition of hospital-associated pathogens and microbial communities by patients during AAI sessions via a multicenter randomized controlled trial; and 3) To determine whether the specific benefits achieved by the visitation program, i.e. reduction in blood pressure, heart rate and self-reported pain and anxiety, are impacted by the interventions. If findings support the hypothesis that chlorhexidine interventions are effective to prevent pathogen transmission through a multicenter, parallel-arm randomized controlled trial and does not reduce Animal-Assisted visitation program benefits to the children or impact the welfare of the therapy dogs, then this will provide strong evidence on which to base recommendations for infection control guidelines for programs nationally.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 3 and 17 years
* Cleared by physician to participate in a hospital-based animal-assisted visitation program session with any enrolled dog

Exclusion Criteria:

* Children who report sensitivity to chlorhexidine products
* Children who report allergy to dogs or sensitivity to dog allergen

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Child MRSA exposure | Baseline through intervention completion, an average of 60 minutes
  MRSA exposure is defined as children who do not have detectable methicillin-resistant Staphylococcus aureus (MRSA) nasal carriage before the dog session who then have MRSA detection (MRSA nasal carriage) after the dog session.

SECONDARY OUTCOMES:
Child Pseudomonas aeruginosa exposure | Baseline through intervention completion, an average of 60 minutes
  Pseudomonas aeruginosa exposure is defined as children who do not have detectable P. aeruginosa nasal carriage before the dog session who then have P. aeruginosa detection after the dog session.
Child and Dog Clostridium difficile prevalence | Baseline to intervention completion, an average of 60 minutes
  Positivity of child and dog for C. difficile at a session

OTHER OUTCOMES:
Dog MRSA fur contamination difference | Baseline through intervention completion, an average of 60 minutes
  Measure of dog dorsal fur ("petting zone") contamination with methicillin-resistant Staphylococcus aureus post session compared to pre session, reported as colony-forming units per dog per visit

CONTACTS AND LOCATIONS:
Overall Officials: Meghan F Davis, DVM, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (3):
- United States (3):
  - Johns Hopkins, Baltimore, Maryland
  - Washington University in St. Louis, St Louis, Missouri
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant meta-data will be linked to microbiome sequencing results and deposited to National Center for Biotechnology Information (NCBI).
Supporting Information: Study Protocol
Time Frame: Data will become available at the time of first publication of the sequencing results.
Access Criteria: There are no specific access criteria instituted by the study. Access will be controlled by NCBI.